CLINICAL TRIAL: NCT01302470
Title: Randomized Study of Endovascular Versus Epicardial Lead Placement for Resynchronization Therapy
Brief Title: Comparison of Epicardial Versus Conventional Lead Placement in Cardiac Resynchronization Therapy
Acronym: REVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-052
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Cardiac Resynchronization Therapy; Heart Failure
Keywords: biventricular pacing
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

ARMS (2):
- Robotic placement of CS lead (Active Comparator): CS leads placed epicardially in the area of increased dyssynchrony as demonstrated by low dose dobutamine stress testing.
  Interventions: Procedure: Primary epicardial placement of left ventricular lead
- Transvenous placement of CS lead (Active Comparator): CS lead will be placed transvenously
  Interventions: Procedure: Transvenous placement of left ventricular lead

INTERVENTIONS:
Procedure: Primary epicardial placement of left ventricular lead — Epicardial leads will be placed on the left ventricle in the area of the most dyssynchrony . the leads will be attached to a Medtronic Cardiac resynchronization/ AICD/ device
  Other Names: cardiac resynchronization therapy
  Arms: Robotic placement of CS lead
Procedure: Transvenous placement of left ventricular lead — Conventional placement of left ventricular leads performed in the electrophysiology department.
  Other Names: Cardiac resynchronization Therapy; CRT/ AICD
  Arms: Transvenous placement of CS lead

SUMMARY:
The primary goal of this study is to evaluate the use of robotically -assisted device leads as a primary strategy for heart resynchronization.This trials aims to compare transvenous lead placement with robotic lead placement for cardiac resynchronization therapy.

DETAILED DESCRIPTION:
A secondary goal is to explore the link between efficacy of CRT and inotropic contractile reserve as measured by dobutamine stress echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic NYHA class III or IV heart failure from idiopathic or ischemic heart failure
* QRS interval greater than or equal to 130 msec
* Left ventricular end diastolic diameter greater than or equal to 55 mm
* left ventricular ejection fraction less than or equal to 35
* Willingness to participate

Exclusion Criteria:

* Acute renal failure; active GI bleeding; unexplained fever which may be due to an infection
* untreated active infection
* acute stroke
* severe uncontrolled systemic hypertension
* severe systemic electrolyte imbalance
* severe concomitant illness that drastically shortens life expectancy
* severe coagulopathy
* history of severe COPD and inability to tolerate single lung ventilation
* History of prior left sided thoracotomy
* history of recent intravenous drug use
* concomitant psychiatric diagnosis that impairs patient's ability to comply with study protocol
* participation in another investigational protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
CHF Hospitalizations & mortality | one year post implant.
  Heart failure and mortality will be assesd along with six minute hall walk tests

CONTACTS AND LOCATIONS:
Locations (1):
- St.Lukes-Roosevelt Hospital, New York, New York, United States